CLINICAL TRIAL: NCT04318249
Title: Behavioral Relaxation Approaches for Insomnia in Lung Cancer Patients
Acronym: LC_ART
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unable to recruit subjects
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Principal Investigator, Nalaka Gooneratne, Principal Investigator, Abramson Cancer Center at Penn Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UPCC 15521; 842655 (Other: University of Pennsylvania IRB)
Record Dates: First submitted 2020-03-18; First posted 2020-03-23 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Insomnia
Keywords: Lung Cancer
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: This will be conducted as a parallel group, single-blinded pilot study for reducing insomnia among lung cancer patients. All subjects will participate in some form of insomnia treatment over a fourteen-day period. Participants eligible and enrolled in the study will be randomized into one of the two arms, which consist of the two different ART. Randomization and survey baseline measurements from eligible participants will occur on day -1 and the intervention period will last until day fourteen. On day thirty, two weeks post intervention(s), surveys will be emailed to participants to track any change in sleep quality, respiratory quality, and perception of sleep.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Assisted Relaxation Therapy (Experimental): This group will be receiving an assisted relaxation therapy intervention
  Interventions: Behavioral: Assisted Relaxation Therapy
- Modified Assisted Relaxation Therapy (Experimental): This group will be receiving a modified version of an assisted relaxation therapy intervention
  Interventions: Behavioral: Assisted Relaxation Therapy; Behavioral: Modified Assisted Relaxation Therapy

INTERVENTIONS:
Behavioral: Assisted Relaxation Therapy — This intervention includes using a smartphone application that helps with breathing techniques and sleep.
Behavioral: Modified Assisted Relaxation Therapy — This intervention includes using a smartphone application that is modified to help with breathing techniques and additional sleep instructions.
  Arms: Modified Assisted Relaxation Therapy

SUMMARY:
This is a randomized, 30-day research study that is exploring the effects of two simplified mindfulness interventions in lung cancer patients aimed to improve their sleep quality and anxiety regarding sleep. The investigators will be enrolling a total of 20 patients who have insomnia symptoms. Patients will use a behavioral intervention to help with their sleep.

DETAILED DESCRIPTION:
The objective is to implement and examine the outcomes of a simplified relaxation intervention, Assisted Relaxation Therapy (ART), for lung cancer patients who experience insomnia symptoms and other sleep difficulties. This intervention includes using a smartphone application. A variety of surveys will be used to track the interventions' efficacy throughout the study. To test these interventions, the investigators will recruit participants (n=20) from a weekly oncology patient list located within the University of Pennsylvania. Participants with a history of lung cancer who are recruited into the study must have a smartphone. Participants will use the ART intervention over the course of 2 weeks and will receive surveys at enrollment (D0), end of intervention (D14) and 2 weeks post-intervention (D30). Missing data will be handled using imputation methods. The investigators will analyze the data using statistical programs to determine progress throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 or older
* Diagnosed with Lung Cancer (In remission, Undergoing Immune Modulated Chemotherapy, Undergoing Platinum-based Chemotherapy
* Fluent in English
* Has Access to Smartphone
* Has internet connection at home
* More than 4 weeks post-surgery

Exclusion Criteria:

* Inability to speak English or communicate verbally
* Medical or other factors that, in the opinion of the study research team, would interfere with their ability to participate in the intervention (such as inability to participate in the guided compassion training due to deafness)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09-30 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Sleep Onset Latency at 14 days | 14 days
  Changes in sleep onset latency will be measured by sleep diary.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No